CLINICAL TRIAL: NCT00190138
Title: Effect of Bi-ventricular Pacing on Autonomous Nervous System
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FEMH-93014; Femh-93-C-014
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-10-07 (Estimated); Status verified 2004-12

CONDITIONS: Congestive Heart Failure
Keywords: Bi-ventricular pacing; ventricular resynchronization; baroreflex sensitivity; heart rate variability
MeSH Terms: conditions — Heart Failure

INTERVENTIONS:
Device: Bi-ventricular pacing

SUMMARY:
Patients with congestive heart failure are often associated with delayed intraventricular depolarization which causing dyssynchrony and an inefficient pattern of left ventricular contraction. A number of studies have shown that bi-ventricular or left ventricular pacing improves indexes of systolic function as well as decreases sympathetic activation in patients with severe left ventricular systolic dysfunction, dilated cardiomyopathy and a major left-sided intraventricular conduction disorder such as left bundle branch block. One recent study also demonstrated that bi-ventricular pacing can shift heart rate variability (HRV) toward a more favorable profile. Baroreflex sensitivity (BRS) is a measure of the negative feedback properties that interact in modulating the dynamic heart rate and arterial pressure fluctuations. Blunted BRS is found to be associated with an increased risk for both cardiac deaths and arrhythmic events. However, the effect of bi-ventricular pacing on BRS has never been studied. In the present proposal, we plan to measure common hemodynamic parameters, BRS and HRV in a group of heart failure patients receiving open heart surgery in different pacing conditions (bi-ventricular pacing, single LV pacing, single RV pacing). The major aims are to investigate the effect of bi-ventricular pacing on BRS and to clarify the underlying mechanisms.

DETAILED DESCRIPTION:
Operation and lead placement:

Off-pump coronary artery bypass (OPCAB) is performed based on patient's coronary angiography. Following the completion of coronary anastomoses, epicardial pacemaker leads are implanted by simple stitches in different locations. The right atrial (RA) lead is placed on the right atrial appendage. The right ventricle (RV) lead is placed on the RV free wall near the apex. The left ventricle (LV) lead is placed on the lateral wall of LV at the border zone between diagonal and obtuse marginal branches of coronary artery. All three ground leads are placed on the rectus abdominis muscle. All these leads are pulled out of the patient percutaneously. Medtronic dual-chamber pacemaker is used for this study. The change of different pacing protocol (RV pacing, LV pacing, or biventricular pacing) is through the connection of different pacemaker leads.

Hemodynamic study:

All patients underwent OPCAB have Swan-Ganz catheter in our institute. Cardiac output measurement is obtained by thermodilution method. Hemodynamic variables (systemic blood pressure, pulmonary artery pressure, central venous pressure, pulmonary capillary wedge pressure, systemic vascular resistance, and pulmonary vascular resistance, etc) are recorded during the measurement.

ECG and blood pressure monitoring system:

ECG and radial arterial blood pressure were recorded by an analog to digital converter system (National Instrument Inc.). The ananlog signals were digitized in a rate of 500Hz and were stored in a hard disk. The data were then analyzed by a program written with MATLAB language (version 5.2, Mathwork Co.). QRS complexes were automatically classified and manually verified as normal sinus rhythm, arterial or ventricular premature beats, or noise by comparison of the adjacent QRS morphologic features. The N-N interval time series were then transferred to a personal computer and post-processed.

Baroreflex sensitivity analysis:

The analysis of BRS was conducted by both the sequence method (19, 20) and the spectral (α-index) method. Sequence method: In brief, the beat-by-beat time series of systolic arterial blood pressure and ECG R-R intervals were scanned to identify sequences of over three consecutive beats in which the systolic blood pressure (SBP) and R-R intervals of the next beat changed concomitantly in increasing or decreasing sequence. Such beat-to-beat sequences were identified as baroreflex sequences. A linear regression was applied to the individual sequence and only r2 values >0.85 were accepted. The measure of each type of the integrated spontaneous BRS was obtained by averaging all accepted slopes of the same type during a 5-minute recording. Spectral (α-index) method: The α-index (α) was obtained by means of the simultaneous spectral analysis of the R-R intervals and the SBP variabilities, with the calculation being made from the square root of the ratio between the R-R intervals and the SBP variability in low frequency (LF) band (αLF, 0.04 to 0.15 Hz). The coherence between the R-R intervals and SBP was assessed by a cross-spectral analysis. The α-index was calculated only when the magnitude of squared coherence (K2) between the RR and the SBP signals exceed 0.5 in LF band.

Heart rate variability analysis:

The missing intervals of the raw N-N data were linearly interpolated and resampled at 4 Hz by the Ron-Berger method. Each 5-minute segment of N-N intervals was taken for HRV analysis. The time domain measurements of HRV included SDNN, r-MSSD. The frequency-domain measurements of HRV included LF and HF, which were calculated by Welch's averaged periodogram of the N-N intervals.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal sinus rhythm proposed to undergo coronary artery bypass surgery.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Kuan-Ming Chiu, M.D., Study Chair — Far Eastern Memorial Hospital